CLINICAL TRIAL: NCT05720104
Title: Effect of Regular Antibacterial Photodynamic Therapy on Oral Hygiene in the Elderly 24-hour Care Residents
Brief Title: Regular Antibacterial Photodynamic Therapy on Oral Hygiene in the Elderly 24-hour Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No new sites have been found to the
Sponsor: Koite Health Oy (Industry)
Collaborators: University of Helsinki (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FlexKoi2022
Record Dates: First submitted 2023-01-19; First posted 2023-02-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Inflamed Gums; Dryness Oral; Plaque
Keywords: Lumoral; Lumorinse; Plaque; Anti-bacterial photodynamic therapy; aPDT; aMMP-8
MeSH Terms: conditions — Gingivitis; Xerostomia; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: Participants in two groups (Study group and Control group) shall receive instructions for standard oral hygiene. The same assessments are done for participants in both groups, and within the same time periods. The Study group will also be using the Lumoral Treatment device.
Masking Description: Participants in two groups (Study group and Control group) shall receive instructions for standard oral hygiene. The same assessments are done for participants in both groups, and within the same time periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Use of Lumoral Treatment device. Standard oral hygiene instructions.
  Interventions: Device: Lumoral Treatment; Other: Standard oral hygiene instructions
- Control group (Other): Standard oral hygiene instructions.
  Interventions: Other: Standard oral hygiene instructions

INTERVENTIONS:
Device: Lumoral Treatment — Subjects will receive detailed instructions for the use of Lumoral treatment -device. Subjects will be instructed to use the Lumoral treatment -device and follow the protocol once a day for two months and to keep a diary.
  Arms: Study group
Other: Standard oral hygiene instructions — Subjects will receive the latest standard oral hygiene instructions according to the Swedish dental association's guidelines.

SUMMARY:
This study aims to determine the effectiveness of the Lumoral device on oral hygiene, inflammatory load, and dryness of mouth in elderly 24-hour care residents. The second aim is to investigate the usefulness and benefits of the aMMP-8 chair-side test and the Lumoral device in improving the oral hygiene of elderly people. In addition, the study will investigate the usability of Lumoral assessed by different care professionals to evaluate the need for oral care and plaque control procedures in elderly residents.

DETAILED DESCRIPTION:
The dental condition of elderly care customers is often poor. Cavities and dental connective tissue disease are widespread in people over 75 and older. Untreated oral infections in patients or residents living in institutional care predispose to pneumonia, among other complications. Chronic oral infectious diseases, and sometimes fatal complications, are preventable with good oral hygiene.

As people get older, their ability to function deteriorates, and the elderly, especially those living in round-the-clock care, have been found to have shortcomings in maintaining oral hygiene. Only a small part of the population had clean teeth, and the worse the level of oral hygiene, the worse the quality of life. Regular cleaning of the mouth and teeth from plaque is still the most important thing for keeping your mouth healthy. Unfortunately, this is not always the case with round-the-clock care, and new practices are needed to improve oral hygiene.

The use of antibacterial photodynamic therapy (aPDT) and antibacterial blue light has been studied and found to reduce the amount of plaque in the mouth. The Lumoral device is a CE-marked home medical device that has been shown to be effective in reducing the development of plaque and harmful bacteria in the plaque. The performance of the device is based on the aPDT method, in which the photosensitive substance in the Lumorinse mouthwash attaches to the bacterial coating and is activated as an antibacterial by light. The antibacterial effect is applied directly to the plaque, reducing the impact on the normal oral flora. Preliminary studies have found that the method reduces inflammatory factors in periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* A 24-hour care resident;
* Understand and able to give consent to the study;
* At least 10 functional teeth in the mouth (including implants);
* Able to brush teeth and follow the instruction for use Lumoral treatment, based on the assessment by the nursing staff.

Exclusion Criteria:

* Incapable of participating in the study based on the assessment of the nursing staff
* Toothless or less than 10 functional teeth in the mouth (including implants)
* Unwilling or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral hygiene | 2 months
  Improvement in oral hygiene / resident experience. The study subject will fill in a questionnaire related to oral hygiene and mouth dryness at baseline and at 2 months.
Visual Plaque Index (VPI) | 2 months
  Change in the Visible plaque index (VPI) is greater in the Study group compared to the Control group.
  VPI:
  * A full-mouth assessment at 4 sites per tooth will be made at baseline and at the 2 month follow-up visit
  * VPI is reported as the percentage (%) of sites with positive findings
  * Dichotomous scoring to each site of the tooth as plaque" 1 present" and" 0 absent"
  * Calculation formula: number of plaque sites/ 4 times number of teeth
Bleeding on Probing (BOP) | 2 months
  Change in the Bleeding on Probing (BOP) is greater in the Study group compared to the Control group.
  BOP:
  * A full-mouth assessment at 4 sites per tooth
  * Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus
  * BOP reported as the percentage (%) of sites with positive findings
  * Dichotomous scoring to each site of the tooth as bleeding" 1 present" and" 0 absent"
  * Calculation formula: number of bleeding sites/ 4 times number of teeth
Probing Pocket Depth (PPD) | 2 months
  Change in the Probing Pocket Depth (PPD) values is greater in the Study group compared to the Control group.
  PPD:
  * A full-mouth assessment, measured at 4 sites per tooth
  * Assessed from the base of the pocket to the gingival margin (mm)
aMMP-8 | 2 months
  Change in the active matrix metalloproteinase 8 values is greater in the Study group compared to the Control group.
  The aMMP-8 marker analysis will be performed using the Periosafe chair-side test (Dentognostics GmbH) according to the manufacturer's instructions.
  Oral rinse samples will be stored for further analysis according to the Swedish Biobanks in Medical Care Act (SFS 2002:297). Further analysis includes aMMP-8 and its regulators by biochemical enzyme/molecule assays, immunoassays, and proteomics analysis.
Dry mouth | 2 months
  Use of the Lumoral Treatment relieves the symptoms of dry mouth, compared to the Control group.
  Clinical assessment of moisture/dryness of oral mucosa (score 0-2) 0 = Saliva secretion looks normal (saliva serous and running)
  1. = Mucous membrane of the mouth shiny and tightening/ saliva foamy or mucous/ little clear saliva at the base of the mouth
  2. = Mouth completely dry, mirror sticking to cheek or tongue, mucous membranes often reddened/ bumps on tongue surface disappeared/ scab on melting

CONTACTS AND LOCATIONS:
Overall Officials: Tommi Pätilä, Docent, Study Director — Koite Health; Timo Sorsa, Professor, Principal Investigator — University of Helsinki
Locations (1):
- Pilträdets servicehus, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Visschere L, de Baat C, De Meyer L, van der Putten GJ, Peeters B, Soderfelt B, Vanobbergen J. The integration of oral health care into day-to-day care in nursing homes: a qualitative study. Gerodontology. 2015 Jun;32(2):115-22. doi: 10.1111/ger.12062. Epub 2013 Jun 20. PMID 23786637
- [Background] Holmen A, Stromberg E, Hagman-Gustafsson ML, Wardh I, Gabre P. Oral status in home-dwelling elderly dependent on moderate or substantial supportive care for daily living: prevalence of edentulous subjects, caries and periodontal disease. Gerodontology. 2012 Jun;29(2):e503-11. doi: 10.1111/j.1741-2358.2011.00507.x. Epub 2011 Sep 19. PMID 21923714
- [Background] Hugoson A, Koch G, Gothberg C, Helkimo AN, Lundin SA, Norderyd O, Sjodin B, Sondell K. Oral health of individuals aged 3-80 years in Jonkoping, Sweden during 30 years (1973-2003). II. Review of clinical and radiographic findings. Swed Dent J. 2005;29(4):139-55. PMID 16463570
- [Background] Lahteenmaki H, Patila T, Raisanen IT, Kankuri E, Tervahartiala T, Sorsa T. Repeated Home-Applied Dual-Light Antibacterial Photodynamic Therapy Can Reduce Plaque Burden, Inflammation, and aMMP-8 in Peri-Implant Disease-A Pilot Study. Curr Issues Mol Biol. 2022 Mar 8;44(3):1273-1283. doi: 10.3390/cimb44030085. PMID 35723308
- [Background] Nikinmaa S, Alapulli H, Auvinen P, Vaara M, Rantala J, Kankuri E, Sorsa T, Meurman J, Patila T. Dual-light photodynamic therapy administered daily provides a sustained antibacterial effect on biofilm and prevents Streptococcus mutans adaptation. PLoS One. 2020 May 6;15(5):e0232775. doi: 10.1371/journal.pone.0232775. eCollection 2020. PMID 32374766
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Nikinmaa S, Podonyi A, Raivio P, Meurman J, Sorsa T, Rantala J, Kankuri E, Tauriainen T, Patila T. Daily Administered Dual-Light Photodynamic Therapy Provides a Sustained Antibacterial Effect on Staphylococcus aureus. Antibiotics (Basel). 2021 Oct 13;10(10):1240. doi: 10.3390/antibiotics10101240. PMID 34680821
- [Background] Nishizawa T, Niikura Y, Akasaka K, Watanabe M, Kurai D, Amano M, Ishii H, Matsushima H, Yamashita N, Takizawa H. Pilot study for risk assessment of aspiration pneumonia based on oral bacteria levels and serum biomarkers. BMC Infect Dis. 2019 Sep 2;19(1):761. doi: 10.1186/s12879-019-4327-2. PMID 31477059
- [Background] Saarela RKT, Hiltunen K, Mantyla P, Pitkala KH. Changes in Institutionalized Older People's Dentition Status in Helsinki, 2003-2017. J Am Geriatr Soc. 2020 Jan;68(1):221-223. doi: 10.1111/jgs.16230. Epub 2019 Oct 26. No abstract available. PMID 31654530
- [Background] Saarela RKT, Hiltunen K, Kautiainen H, Roitto HM, Mantyla P, Pitkala KH. Oral hygiene and health-related quality of life in institutionalized older people. Eur Geriatr Med. 2022 Feb;13(1):213-220. doi: 10.1007/s41999-021-00547-8. Epub 2021 Jul 27. PMID 34313976
- [Background] Suominen AL, Varsio S, Helminen S, Nordblad A, Lahti S, Knuuttila M. Dental and periodontal health in Finnish adults in 2000 and 2011. Acta Odontol Scand. 2018 Jul;76(5):305-313. doi: 10.1080/00016357.2018.1451653. Epub 2018 Mar 16. PMID 29546776
- [Background] Willumsen T, Karlsen L, Naess R, Bjorntvedt S. Are the barriers to good oral hygiene in nursing homes within the nurses or the patients? Gerodontology. 2012 Jun;29(2):e748-55. doi: 10.1111/j.1741-2358.2011.00554.x. Epub 2011 Oct 24. PMID 22023222
- See also: Alaijah, F., Morsi, A., Nasher, R. et al. Photobiomodulation therapy in the treatment of periodontal disease: a literature review. Laser Dent Sci 3, 147-153 (2019) — https://link.springer.com/article/10.1007/s41547-019-00056-9
- See also: Levine JI (1990). Medications that increase photosensititivity. FDA document Dec 1990. — https://www.fda.gov/media/75892/download
- See also: United Nations Population Division. World Population Prospects: The 2002 Revision. New York, NY, USA: United Nations, 2003. — https://www.un.org/development/desa/pd/sites/www.un.org.development.desa.pd/files/files/documents/2020/Jan/un_2002_world_population_prospects-2002_revision_volume-ii.pdf